CLINICAL TRIAL: NCT06436131
Title: The Effects of In-phase Bilateral Exercise on Cognitive and Motor Outcome Measures, in Patients with Progressive Multiple Sclerosis, a Randomized Control Trial.
Brief Title: The Effects of In-phase Bilateral Exercise in People with Progressive Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: Cyprus Institute of Neurology and Genetics (Other)
Responsible Party: Principal Investigator, Dimitris Sokratous, Principal Investigator, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IBEPMS
Record Dates: First submitted 2024-03-19; First posted 2024-05-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive
Keywords: In-phase Bilateral; exercise; cognitive processing; multiple sclerosis; manual dexterity
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Motor Activity; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Subjects were randomized in two groups. Experimental group received an exercise program based on in-phase bilateral exercises, whereas the active control group receives conservative exercises. The duration of the study was 12 consecutive weeks for both groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: It was a double-blind study in which neither the participants nor the assessor and the trainer knew who's been assigned to either group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IBPMS (Experimental): The exercise program of the experimental group consisted of exercises based on in-phase bilateral movements of the upper and lower limbs, which they were adapted to different sport activities and to fitness functional exercises. The specific exercise program was organized in a group circuit training, performed simultaneously on each session from all the participants of the experimental group, considering the MS exercise recommendations. Specifically, the program included sports activities of basic technical skills of basketball (e.g., different types of passing, catching and throwing the ball) and volleyball (e.g., different types of passing and receiving the ball), whereas the fitness exercises included the diagonal movements from proprioceptive neuromuscular facilitation technique, by the use of a resistance bands.
  Interventions: Behavioral: In-phase Bilateral Exercise
- Controls (Active Comparator): The participants of the active control group, underwent an exercise program based on conventional exercises, such as strengthening of the major muscle groups of the trunk, resistance exercises for the upper and lower limbs and body weight support treadmill exercise. All participants of the active control group performed the specific types of exercises individually, as opposed with the experimental group which was organized as a group training. Controls performed the specific type exercises once a week, for 12 consecutive weeks.
  Interventions: Behavioral: Conservative exercises

INTERVENTIONS:
Behavioral: In-phase Bilateral Exercise — The exercise program of the experimental group consisted of exercises based on in-phase bilateral movements of the upper and lower limbs, which were adapted to different sport activities and to fitness functional exercises.
  The participants of experimental group performed the specific type exercises three times per week, for 12 consecutive weeks.
  Arms: IBPMS
Behavioral: Conservative exercises — The participants of the active control group, underwent an exercise program based on conventional exercises, such as strengthening of the major muscle groups of the trunk, resistance exercises for the upper and lower limbs and body weight support treadmill exercise.
  Arms: Controls

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the central nervous system. MS, typical presents with progression of clinical symptoms which mainly include motor and cognitive impairment, as well as reduction of patients' quality of life. Exercise is an effective approach in the management of the symptoms in people with progressive MS. Previous studies in healthy and in people with MS, reported a close relationship between cognitive functions and upper limb performance. Since patients with progressive MS facing difficulties with performing complex exercises due to cognitive dysfunctions and given the close relationship between cognitive functions and manual dexterity, a reasonable question arises whether a type of upper limbs exercises with less cognitive demands will improve the information processing speed in people with progressive MS. The aim of the current study is to investigate the effects of in-phase bilateral upper limbs exercises on the information processing speed, in patients with progressive MS, given that in-phase bilateral movements needs less attentional load than the other types of bilateral coordination. The intervention protocol lasted for 12 consecutive weeks (30-60 minutes /session x 3 sessions/week) and included in-phase bilateral exercises of the upper limbs, adapted to different sports activities and to functional training. Results from the statistical analysis indicated improvement of the experimental group compared to the control group, on the information processing speed alongside with improvement of motor skills.

DETAILED DESCRIPTION:
The term progressive multiple sclerosis (MS) includes both secondary progressive MS (SPMS) and primary progressive MS (PPMS). As it is well known, the course of MS is highly variable. On one hand, almost 50% of the patients who is characterized by the relapsing remitting MS, after 10-15 years of disease this pattern becomes progressive, in which individual clinical symptoms slowly progress, a disease type defined as a SPMS. On the other hand, in about 15% of people with MS, disease progression is persistent from onset defined as a PPMS. Patients with progressive MS except from physical impairment, often have cognitive dysfunctions, which negatively affect quality of life. Information processing speed is the most common cognitive deficit, between people with PPMS and those with SPMS.

Despite the fact that cognitive rehabilitation approaches are effective in treating MS-related cognitive dysfunctions, there are evidence from several studies which indicated the impact of different types of exercises in the improvement of cognitive in people with MS. Furthermore, evidences from previous studies in healthy and people with MS, reported a close relationship between cognitive functions and upper limbs performance, defined by the projections from the Anterior Cingulate Cortex to the motor cortex and spinal cord. Specifically, the decline of information processing speed indicates reduction of manual dexterity in people with MS. Manual dexterity is defined as the manual skill which contains coordination of fine and gross voluntary movements of the upper limbs. Manual dexterity dysfunction in MS contributes to reduced ability to perform activities of daily living (ADLs) and social activities, which causes reduction of independency and quality of life.

Moreover, evidence from previous studies, reported that in-phase bilateral movements needs less attentional load and less neural control than the unilateral or the other types of bilateral coordination, as a result to perform the specific type of movement (i.e., in-phase bilateral) more efficient and more easy. Therefore, given that patients with progressive MS characterized by decline of information processing speed, which affects manual dexterity, a reasonable question arises whether in-phase bilateral upper limbs exercises will improve information processing speed and thus, to improve manual dexterity in the specific clinical cohort.

The aim of the current study was to investigate primarily the hypothesis that a 12-week exercise program based on in-phase bilateral upper limbs movements, based on sport activities and functional training, could improve information processing speed compared to a conservative type of exercise, in people with progressive MS. A secondary aim was to evaluate whether the specific exercise program could improve manual dexterity and have a correlation with information processing speed.

Second aim of the study was to investigate the effects of the specific type of exercises on various clinical symptoms, fatigue and on quality of life, using clinical assessment tools and subjective questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of progressive multiple sclerosis (MS) (primary or/and secondary progressive MS)
* Expanded Disability Status Scale score between three and six
* no relapse within 30 days
* aged between 30 and 70 years
* Mini Mental State of Examination score between 20 and 30 (mild to no cognitive impairment)

Exclusion Criteria:

* history of any disease affecting the central nervous system other than MS (e.g., stroke, Parkinson's disease, cerebral palsy)
* history of cardiovascular disease (e.g., known aneurism, myocardial infarction, hyper/hypotension, heart failure)
* severe orthopaedic disorders (e.g., knee or hip replacement, spondylosurgery, disk herniation, recent bone fracture)
* mental disorders (e.g., depression, schizophrenia, bipolar syndrome)
* pregnancy during the implementation of the study timeline
* hearing impairments (i.e., deafness)
* visual deficit (e.g., optic neuritis, blindness, diplopia, glaucoma, blurred vision)
* history of epileptic seizures
* spasticity level on upper or lower limbs more than 1+ (slight increase in muscle tone) according to Modified Ashworth Scale

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test | Baseline (3 weeks) until the end of the Intervention (12 weeks)
  It is a commonly used test in pwMS, which measures processing speed as well as motor speed. The investigators employed the oral form of the test, in which participants were provided with the test sheet with nine symbols, each paired with a number on top of the page, defined as the "key". For example, the symbol "O" is matched with the number "6", so the correct response would be "six". The rest of the page consists of a randomized, sequential variety of these symbols. Participants are asked to verbally respond with the number that corresponds with each symbol. During the test, the participant is given two minutes to orally match symbols with digits as quickly as possible. The score is obtained by subtracting the number of errors from the number of items completed. To account for practice effects, the investigators created six different tests, as many as our assessment points, in which the order of the symbols and the numbers of the "key" were rearranged

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form 36 | Baseline (3rd week) until the end of the Intervention (12 weeks)
  It is a set of generic, coherent, and easily administered quality-of-life measures, completed by the participants. There are 11 questions in the specific questionnaire administered by an assessor, with 36 items in total, which cover eight domains scaled from 0 to 100, with higher values indicating better health status. The eight domains include: general health, vitality, physical function, role physical, bodily pain, role emotional, social functioning and mental health. It takes between 5 and 10 min to complete it.
Modified Fatigue Impact Scale | Baseline (3rd week) until the end of the Intervention (12 weeks)
  It is a short questionnaire which requires the participants to describe the effects of fatigue during the past four weeks. The Modified Fatigue Impact Scale consists of 21 questions which are subjectively rated from "0" (low rate) to "4" (high rate) and it is divided into three subscales (i.e., physical, cognitive, and psychosocial). The assessor records the total score of the test as the final test result. The higher the score is, the greater is the impact of fatigue in individual daily life. Therefore, the Modified Fatigue Impact Scale it is used as the description of participants' attribution of functional restrictions to fatigue symptoms.
Trail Making Test | Baseline (3 weeks) until the end of the Intervention (12 weeks)
  It contains five conditions; the visual scanning, motor speed, number sequencing, letter sequencing, and number-letter switching. Trail Making Test also assesses attention, information processing speed and mental flexibility. This particular test consists of two parts, A and B, which involves 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the participant should connect the numbers in ascending order by drawing lines. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the participants connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (e.g., 1-A-2-B-3-C, etc.). The participants were instructed to connect the circles as quickly as possible, without lifting the pencil from the paper. During participants' connection of the "trails", the assessor notes possible errors, and the time needed to complete the task.
Purdue Pegboard Test | Baseline (3 weeks) until the end of the Intervention (12 weeks)
  It is a standardized test of manual dexterity. The Purdue Pegboard Test consists of four subtests, performed in a board in which pins, washers and collars are placed by the participants into two parallel columns of holes, according to the subtest task. The first two subtests are unimanual tasks, which measure dexterity of the right and left hand, respectively. The third subtest is a synchronous bimanual task that requires simultaneous use of both hands to grasp pins and place them in their corresponding columns of holes. During the fourth subtest, the participants should perform alternating movements of both hands to complete assemblies of different types of pegs. Standard scoring of the Purdue Pegboard Test is based on the number of pegs inserted in 30 s for the first three subtests, and in 1 min for the last subtest.
Timed 25-Foot Walk | Baseline (3 weeks) until the end of the Intervention (12 weeks)
  It is a quantitative assessment for mobility and lower limb function. Participants are directed to one end of a marked 25-foot path and they are instructed to walk as quickly as possible. The time is recorded from the start and ended when participants reached the 25-foot mark. The same task is immediately run again by having the participants walked back the same distance. Due to the fact that our participants might be using assistive devices for walking, they are instructed to use them in order to be safe when doing this task. The final score for each participant, is the mean score from the two completed trials.
Six Spot Step Test | Baseline (3 weeks) until the end of the Intervention (12 weeks)
  It is a measure replicating a complex range of sensorimotor functions, such as lower limb strength, spasticity, coordination, as well as balance. It is a timed walking test that involves kicking over a number of targets placed along a 5 meter path. The specific test is cognitive demanding, that also includes coordination and dynamic balance.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Sokratous, Principal Investigator — Cyprus University of Technology
Locations (1):
- Dimitris Sokratous, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
The data from the two study groups will be available in figshare repository.
Supporting Information: Study Protocol, SAP
Time Frame: When summary data are published then all Data will be available
Access Criteria: Raw data will available for any scientist who wants to analyze or for reproducibility

REFERENCES:
- [Background] DeLuca J, Chiaravalloti ND, Sandroff BM. Treatment and management of cognitive dysfunction in patients with multiple sclerosis. Nat Rev Neurol. 2020 Jun;16(6):319-332. doi: 10.1038/s41582-020-0355-1. Epub 2020 May 5. PMID 32372033
- [Background] Bush G, Luu P, Posner MI. Cognitive and emotional influences in anterior cingulate cortex. Trends Cogn Sci. 2000 Jun;4(6):215-222. doi: 10.1016/s1364-6613(00)01483-2. PMID 10827444
- [Background] Paus T. Primate anterior cingulate cortex: where motor control, drive and cognition interface. Nat Rev Neurosci. 2001 Jun;2(6):417-24. doi: 10.1038/35077500. PMID 11389475
- [Background] Grefkes C, Eickhoff SB, Nowak DA, Dafotakis M, Fink GR. Dynamic intra- and interhemispheric interactions during unilateral and bilateral hand movements assessed with fMRI and DCM. Neuroimage. 2008 Jul 15;41(4):1382-94. doi: 10.1016/j.neuroimage.2008.03.048. Epub 2008 Apr 8. PMID 18486490
- [Background] Swinnen SP, Wenderoth N. Two hands, one brain: cognitive neuroscience of bimanual skill. Trends Cogn Sci. 2004 Jan;8(1):18-25. doi: 10.1016/j.tics.2003.10.017. PMID 14697399
- [Background] Sokratous D, Charalambous CC, Papanicolaou EZ, Michailidou K, Konstantinou N. Investigation of in-phase bilateral exercise effects on corticospinal plasticity in relapsing remitting multiple sclerosis: A registered report single-case concurrent multiple baseline design across five subjects. PLoS One. 2023 Mar 2;18(3):e0272114. doi: 10.1371/journal.pone.0272114. eCollection 2023. PMID 36862693